CLINICAL TRIAL: NCT00066612
Title: Phase II Study of Irinotecan in Patients With Advanced Transitional Cell Carcinoma of the Urothelium
Brief Title: S0306, Irinotecan in Treating Patients With Recurrent or Refractory Advanced Transitional Cell Cancer of the Urothelium Previously Treated With Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000316428; U10CA032102 (NIH); S0306 (Other: SWOG)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: recurrent bladder cancer; stage IV bladder cancer; metastatic transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter; transitional cell carcinoma of the bladder; anterior urethral cancer; posterior urethral cancer; recurrent urethral cancer; urethral cancer associated with invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Irinotecan
  Interventions: Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: irinotecan hydrochloride — Irinotecan will be given 250 mg/m^2 through intravenous (IV) for 90 minutes on day 1 for every 21 days until tumor progression or unacceptable toxicity or other reason for discontinuation occurs

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as irinotecan use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irinotecan in treating patients who have recurrent or refractory advanced transitional cell cancer of the urothelium.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the probability of response (confirmed complete and partial response) to treatment with irinotecan in patients with recurrent or refractory advanced transitional cell carcinoma of the urothelium previously treated with platinum-based chemotherapy.
* Determine the qualitative and quantitative toxic effects of this drug in these patients.
* Determine the overall and progression-free survival of patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to prior pelvic radiotherapy (yes vs no).

Patients receive irinotecan IV over 90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 5-10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell carcinoma (TCC) of the urothelium, including the bladder, renal pelvis, ureter, and urethra

  * Stage T2-4, N0-3, M1 OR stage T2-4, N+, M0, unresectable disease
  * The following additional histologic subtypes are eligible:

    * Poorly differentiated TCC
    * Predominant TCC with rare foci of squamous differentiation
    * Predominant TCC with rare foci of adenocarcinoma
  * The following histologic subtypes are ineligible:

    * Adenocarcinoma
    * Small cell carcinoma
    * Sarcoma
    * Squamous cell carcinoma
    * Mixed adeno/squamous/transitional histology
* Incurable by surgery or radiotherapy
* Progressed or recurred after 1, and only 1, prior cisplatin- or carboplatin-containing systemic regimen for metastatic disease
* Measurable disease

  * Soft tissue disease that has been irradiated within the past 2 months is not considered measurable disease
* No uncontrolled central nervous system (CNS) metastases

  * CNS metastases that have responded to or stabilized after prior radiotherapy are allowed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count at least 1,200/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (SGOT) less than 3 times ULN (5 times ULN if liver metastases are present)

Renal

* Creatinine less than 2 times ULN

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer that is currently in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* At least 28 days since prior chemotherapy
* No prior topoisomerase I inhibitors (e.g., irinotecan or topotecan)

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 28 days since prior radiotherapy to the pelvis

Surgery

* Not specified

Other

* Recovered from prior therapy
* Prior adjuvant therapy allowed
* At least 14 days since prior Hypericum perforatum (St. John's Wort)
* More than 7 days since prior phenytoin, phenobarbital, carbamazepine, or any other enzyme-inducing anticonvulsant drugs (EIACDs)
* No St. John's Wort during and for 7 days after study participation
* No concurrent EIACDs
* No concurrent medications that cause myelosuppression
* No concurrent medications that cause diarrhea
* Concurrent gabapentin or other non-EIACDs are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-07; Primary Completion 2007-08 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Probability of response (confirmed complete and partial response) | From date of registration to date of progression or death from any cause, whichever came first, assessed up to 3 years

SECONDARY OUTCOMES:
Number and grade of adverse events | From date of registration to date of progression or death from any cause, whichever came first, assessed up to 3 years
Overall survival | From date of registration to date of progression or death from any cause, whichever came first, assessed up to 3 years
Progression-free survival | From date of registration to date of progression or death from any cause, whichever came first, assessed up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz M. Beer, MD, Study Chair — OHSU Knight Cancer Institute

REFERENCES:
- [Result] Beer TM, Goldman B, Nichols CR, Petrylak DP, Agarwal M, Ryan CW, Crawford ED; Southwest Oncology Group. Southwest Oncology Group phase II study of irinotecan in patients with advanced transitional cell carcinoma of the urothelium that progressed after platinum-based chemotherapy. Clin Genitourin Cancer. 2008 Mar;6(1):36-9. doi: 10.3816/cgc.2008.n.006. PMID 18501081